CLINICAL TRIAL: NCT05609578
Title: A Phase 2 Trial of Combination Therapies With Adagrasib in Patients With Advanced Non-Small Cell Lung Cancer With KRAS G12C Mutation
Brief Title: Combination Therapies With Adagrasib in Patients With Advanced NSCLC With KRAS G12C Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0010; 849-017 (Other: Mirati Therapeutics Protocol ID); CA239-0010 (Other: Bristol-Myers Squibb Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Advanced NSCLC; Metastatic Lung Cancer
Keywords: KRAS G12C; NSCLC; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: PD-L1 TPS≥ 1% (Closed) (Experimental): Adagrasib 400 mg BID for 2 cycles followed by adagrasib 400 mg BID + pembrolizumab 200 mg every 3 weeks (Q3W) up to 35 cycles
  Interventions: Drug: Adagrasib oral dose of 400 mg twice daily tablets
- Cohort C (Experimental): Adagrasib 400 mg BID + pemetrexed 500 mg/m2 Q3W + pembrolizumab 200 mg Q3W up to 31 cycles
  Interventions: Drug: Adagrasib oral dose of 400 mg twice daily tablets; Combination Product: Pembrolizumab; Combination Product: Chemotherapy: Pemetrexed; Combination Product: Cisplatin/Carboplatin
- Cohort E (Experimental): Adagrasib 400 mg BID + pembrolizumab 200 mg Q3W + pemetrexed 500 mg/m2 + cisplatin 75 mg/m2 Q3W OR carboplatin AUC 5 Q3W for 4 cycles, followed by adagrasib 400 mg BID + pemetrexed 500 mg/m2 Q3W + pembrolizumab 200 mg Q3W (up to 31 cycles)
  Interventions: Drug: Adagrasib oral dose of 400 mg twice daily tablets; Combination Product: Pembrolizumab; Combination Product: Chemotherapy: Pemetrexed; Combination Product: Cisplatin/Carboplatin

INTERVENTIONS:
Drug: Adagrasib oral dose of 400 mg twice daily tablets — oral dose of 400 mg twice daily tablets
Combination Product: Pembrolizumab — IV infusion once every 3 weeks
  Arms: Cohort C; Cohort E
Combination Product: Chemotherapy: Pemetrexed — IV infusion once every 3 weeks
  Arms: Cohort C; Cohort E
Combination Product: Cisplatin/Carboplatin — IV infusion once every 3 weeks
  Arms: Cohort C; Cohort E

SUMMARY:
Study CA239-0010 is an open-label, Phase 2 clinical trial evaluating the clinical efficacy of adagrasib in combination with pembrolizumab and chemotherapy in the first-line setting for patients with advanced NSCLC with TPS ≥ 1%, TPS <50% and KRAS G12C mutation

ELIGIBILITY:
Cohort A* (closed): Has an untreated and unresectable or metastatic NSCLC with histologically confirmed (squamous or nonsquamous) KRASG12C mutation and histologically confirmed PD-L1 TPS ≥1%.

* Cohort C: Has an untreated and unresectable or metastatic NSCLC with histologically confirmed (non-squamous only) KRASG12C mutation and histologically confirmed PD-L1 TPS < 50% AND previously completed 4 cycles of standard-of-care platinum based induction chemotherapy with pembrolizumab AND experienced stable disease, partial response, or complete response per investigator's assessment after 4 cycles OR if patients received <4 cycles of a platinum-based induction, was stopped early due to intolerable toxicity
* Cohort E: Has an untreated and unresectable or metastatic NSCLC with histologically confirmed (non-squamous only) KRASG12C mutation and histologically confirmed PD-L1 TPS < 50%
* Presence of measurable disease per RECIST v1.1

Exclusion Criteria:

* All Cohorts: Any prior therapy targeting KRASG12C mutation in any setting
* Cohorts A & E: Prior systemic therapy for locally advanced or metastatic NSCLC, including chemotherapy, immune checkpoint inhibitor therapy or chemoimmunotherapy (note: prior systemic therapy or chemoradiation given in the adjuvant or neoadjuvant setting are allowed if last dose of prior systemic treatment was >1 year prior to first dose of study treatment)
* Cohort C: received maintenance therapy (e.g, pembrolizumab and/or pemetrexed following completion of 4-6 cycles of a platinum-based regimen administered in the first-line setting
* Radiation to the lung > 30 Gy within 6 months prior to first dose of study treatment
* Active brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) for Cohort A and E | 30 months
  Defined as the percent of patients documented to have a confirmed CR or PR
Progression-free Survival (PFS) at six months for Cohort C | 30 months
  PFS is defined as time from first study treatment until disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse Events | 30 months
  Defined as number of patients with treatment emergent AEs
Duration of Response (DOR) | 30 months
  Defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of either Progression of Disease (PD) or death due to any cause, whichever occurs first.
Overall Survival (OS) | 30 months
  Defined as time from date of first study treatment to date of death due to any cause
Progression-free Survival (PFS) | 30 months
  Defined as time from first study treatment until disease progression or death from any cause, whichever occurs first.
Population pharmacokinetic (PK) Model Derived AUC at Steady State (AUCtau,ss). | Time Frame: Pre-dose and 4-6 hours post dose; up to 6 months
  Concentration data from this study will be pooled with other studies and exposure parameters derived using population PK methods. Data for this Outcome Measure will not be reported here since ClinicalTrials.gov is designed to report results from participants enrolled in the study and described in the Participant Flow module.
Cohorts C and E: DLTs during SLI (Safety Lead In) | 30 months
  Defined as those patients in the SLI of the study who have received at least 80% of the assigned dose of adagrasib during the first cycle on study, or interrupted or discontinued study treatment during the first cycle due to a DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (166):
- United States (84):
  - Local Institution - Unk025, Anchorage, Alaska
  - Local Institution - 017-591, Glendale, Arizona
  - Local Institution - 017-821, Phoenix, Arizona
  - Local Institution - Unk047, Anaheim, California
  - Local Institution - 017-936C, Fountain Valley, California
  - MemorialCare - Orange Coast Medical Center, Fountain Valley, California
  - Providence Medical Foundation - Virginia K. Crosson Cancer Center - Fullerton, Fullerton, California
  - Local Institution - Unk004, Loma Linda, California
  - Local Institution - 017-961, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Local Institution - 017-872-I, Aurora, Colorado
  - Local Institution - 017-872-G, Boulder, Colorado
  - Local Institution - 017-872-D, Colorado Springs, Colorado
  - Local Institution - 017-872-J, Colorado Springs, Colorado
  - Local Institution - 017-872-B, Denver, Colorado
  - Local Institution - 017-872-F, Denver, Colorado
  - Local Institution - 017-872-A, Lakewood, Colorado
  - Local Institution - 017-872-C, Littleton, Colorado
  - USOR - Rocky Mountain Cancer Centers - Lone Tree - Sky Ridge Medical Center, Lone Tree, Colorado
  - Local Institution - 017-872-E, Pueblo, Colorado
  - Local Institution - 017-872-H, Thornton, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - The Oncology Institute of Hope and Innovation - Lakeland, Lakeland, Florida
  - Local Institution - Unk076, Miami, Florida
  - Local Institution - Unk055, Orlando, Florida
  - Local Institution - Unk062, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Local Institution - 017-820J, Fairway, Kansas
  - Local Institution - 017-820A, Kansas City, Kansas
  - Local Institution - 017-820B, Kansas City, Kansas
  - Local Institution - 017-820C, Kansas City, Kansas
  - Local Institution - 017-820H, Kansas City, Kansas
  - Local Institution - 017-820I, Overland Park, Kansas
  - University of Kansas Cancer Center - Westwood/Richard and Annette Bloch Cancer Care Pavilion, Westwood, Kansas
  - Local Institution - 017-965, Lexington, Kentucky
  - Local Institution - Unk009, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - Unk039, Burlington, Massachusetts
  - Local Institution - Unk069, Detroit, Michigan
  - Local Institution - Unk018, Lansing, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Local Institution - 017-838B, Minneapolis, Minnesota
  - Local Institution - 017-838C, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium (MMCORC), Saint Louis Park, Minnesota
  - Local Institution - 017-838A, Saint Louis Park, Minnesota
  - Local Institution - 017-820F, Kansas City, Missouri
  - Local Institution - 017-820E, Kansas City, Missouri
  - Local Institution - 017-820D, Lee's Summit, Missouri
  - Local Institution - 017-820G, North Kansas City, Missouri
  - Local Institution - Unk008, Osage Beach, Missouri
  - Local Institution - Unk058, Springfield, Missouri
  - Local Institution - 017-080, Babylon, New York
  - Local Institution - 017-088, Brooklyn, New York
  - Hematology-Oncology Associates of Central New York - Brittonfield - East Syracuse, East Syracuse, New York
  - Local Institution - 017-087, New Hyde Park, New York
  - Local Institution - 017-085, New York, New York
  - Local Institution - 017-082, Patchogue, New York
  - Local Institution - 017-086, Port Jefferson, New York
  - Local Institution - 017-081, Port Jefferson Station, New York
  - New York Cancer & Blood Specialists - Cancer Center - Research Headquarters, Port Jefferson Station, New York
  - Local Institution - 017-084, Riverhead, New York
  - Local Institution - 017-945, The Bronx, New York
  - Local Institution - 017-083, The Bronx, New York
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Local Institution - 017-836, Kettering, Ohio
  - Local Institution - 017-916, Memphis, Tennessee
  - Texas Oncology - Dallas Fort Worth (DFW) - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Local Institution - Unk056, Dallas, Texas
  - Local Institution - 017-848, Houston, Texas
  - Local Institution - 017-999, Irving, Texas
  - USOR - Texas Oncology Northeast Texas - Longview Cancer Center, Longview, Texas
  - Local Institution - 017-878-B, Palestine, Texas
  - Local Institution - 017-878-C, Paris, Texas
  - Local Institution - 017-878-A, Tyler, Texas
  - Local Institution - Unk010, Salt Lake City, Utah
  - Local Institution - 017-814-A, Arlington, Virginia
  - Local Institution - Unk066, Fairfax, Virginia
  - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
  - Local Institution - 017-814-B, Gainesville, Virginia
  - Local Institution - 017-814-C, Reston, Virginia
  - PeaceHealth St. Joseph Medical Center, Bellingham, Washington
  - Local Institution - Unk036, Huntington, West Virginia
- Brazil (9):
  - Local Institution - 017-458, Natal, Rio Grande do Norte
  - Local Institution - 017-446, Ijuí, Rio Grande do Sul
  - Local Institution - 017-453, Itajaí, Santa Catarina
  - Local Institution - 017-457, Barretos
  - Local Institution - 017-442, Curitiba
  - Local Institution - 017-452, Fortaleza
  - Local Institution - 017-455, Jaú
  - Local Institution - 017-454, Rio de Janeiro
  - Local Institution - 017-456, São Paulo
- Chile (4):
  - Local Institution - 017-695, Viña del Mar, Región de Valparaíso
  - Local Institution - 017-697, Providencia
  - Local Institution - 017-696, Santiago
  - Local Institution - 017-698, Temuco
- France (17):
  - Institut de Cancerologie de lOuest - Angers, Angers
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Georges Francois Leclerc, Dijon
  - Hopital Michallon, La Tronche
  - Local Institution - 017-688, Lille
  - Local Institution - Unk078, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Local Institution - Unk067, Marseille
  - Local Institution - 017-200, Montpellier
  - Local Institution - Unk029, Paris
  - Hopital Tenon, Paris
  - Local Institution - 017-664, Paris
  - Local Institution - 017-198, Saint-Herblain
  - Hopital Foch, Suresnes
  - Hopital Larrey, Toulouse
  - Gustave Roussy, Villejuif
- Georgia (6):
  - Local Institution - 017-790, Batumi
  - Local Institution - 017-789, Tbilisi
  - Local Institution - 017-794, Tbilisi
  - Local Institution - 017-791, Tbilisi
  - Local Institution - 017-792, Tbilisi
  - Local Institution - 017-793, Tbilisi
- Greece (3):
  - University General Hospital of Heraklion (PAGNI), Heraklion
  - University General Hospital of Larissa, Larissa
  - Metropolitan Hospital, Piraeus
- Hungary (4):
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Italy (12):
  - Local Institution - 017-767 - B, Faenza, Ravenna
  - Local Institution - 017-767 - A, Lugo, Ravenna
  - Azienda Ospedaliera San Giuseppe Moscati - Avellino, Avellino
  - Local Institution - 017-274, Aviano
  - Ospedale Santo Spirito, Casale Monferrato
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano
  - Local Institution - 017-297, Padua
  - Ospedale Santa Maria delle Croci di Ravenna, Ravenna
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma
  - Local Institution - 017-280, Roma
- Malaysia (4):
  - Local Institution - 017-076, Kota Bharu, Kelantan
  - Local Institution - 017-075, Kuantan, Pahang
  - Local Institution - 017-073, Kuala Lumpur
  - Local Institution - 017-072, Putrajaya
- Poland (4):
  - Local Institution - 017-381, Konin
  - Instytut MSF, Lodz
  - Med Polonia Sp. z o. o. - Obornicka, Poznan
  - Wojskowy Instytut Medyczny, Warsaw
- Serbia (5):
  - Local Institution - 017-692, Belgrade
  - Local Institution - 017-693, Belgrade
  - Local Institution - 017-690, Belgrade
  - Local Institution - 017-691, Kamenitz
  - Local Institution - 017-694, Kragujevac
- Spain (9):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Local Institution - Unk001, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Local Institution - 017-395, Geneva, Switzerland
- Thailand (4):
  - Local Institution - 017-132, Bang Phlat
  - Local Institution - 017-136, Bangkok
  - Local Institution - 017-135, Chom Thong
  - Local Institution - 017-137, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05609578.html